CLINICAL TRIAL: NCT00145743
Title: Diagnostics and Therapy of Disease-Related Quality of Life of Patients With Breast Cancer: Protocol of a Randomized Clinical Trial at the Tumor Center Regensburg
Brief Title: Diagnostics and Therapy of Disease-Related Quality of Life of Patients With Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tumor Center Regensburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUZ-QL-RS-04; 3.5/8203-1/117/02
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Breast Neoplasms
Keywords: Quality of Life; Breast Cancer; Referee's Report; Diagnostics; Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patient's reported questionaire, profile in 10 dimensions (EORTC) and referees' report with treatment recommendations
  Interventions: Behavioral: physio,pain,psychotherapy;social,nutrit.counselling&sports
- 2 (Experimental): Patient's reported questionaire; no recommendations given
  Interventions: Behavioral: physio,pain,psychotherapy;social,nutrit.counselling&sports

INTERVENTIONS:
Behavioral: physio,pain,psychotherapy;social,nutrit.counselling&sports — profile and treatment recommendations based on the profile vs. routine psychooncology

SUMMARY:
Quality of Life-Diagnostics and -Therapy in Individual Patients with Breast Cancer.

A randomized study including 200 patients, 5 clinics and 43 general practitioners as coordinating doctors for quality of life therapies.

DETAILED DESCRIPTION:
Quality of life (QL) is increasingly being accepted as an important endpoint in clinical studies, however little is known about its diagnostic value in order to optimize the therapy of cancer patients. This project at the Tumorcentre Regensburg aims to integrate QL-diagnostics into the therapy of patients with breast cancer and to evaluate the efficacy of QL-diagnostics in the context of a randomized clinical trial.

The Tumorcentre Regensburg provides the infrastructure of the present project (telemedicine, project groups, quality circle). Breast cancer patients' therapy is based on the recent national breast cancer therapy guideline, including assorted QL-enhancing therapy options, such as pain therapy, physiotherapy and lymphatic drainage, psychotherapy, social counseling and rehabilitation, nutrition and sports.

In the course of an implementation phase, a new method of QL diagnostics has been developed. Five experts with varying professional background use the individual patient's QL profile and clinical and sociodemographic information in order to generate a QL-report including a therapy recommendation.

This is a two-arm randomized clinical trial with one test group (communication of the QL-finding to the coordinating physician) and a control group (no communication). Patients with newly diagnosed breast cancer who are treated in the study region by one of the coordinating doctors will be included in this randomized study. QL-assessments (EORTC QLQ-C30 plus BR23) will be taken at designated points in time over a 12 months time course. Finally, patients will provide an overall evaluation of the course and the effects of the therapy using an open-ended questionnaire.

We expect that patients in the test group will experience a lower number of QL-deficits at the end of the study period (Median 1 +/- 2) than patients of the control group (Median 2 +/- 2). The statistical confirmation of this expected effect requires a total sample size of N = 200 (n=100 vs. n=100, alpha = 5% [two-tailed], beta = 10%).

This is the first study to evaluate a new form of QL-diagnostics in the complexity of a real patient care environment. This study promises to reveal important new insights into advanced patient care and will make the inclusion of the quality of life concept in the current breast cancer treatment guideline more concrete.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary breast cancer in the county of Regensburg, Amberg and Sulzbach-Rosenberg from November 2004 to approximately June 2006 submitted by coordinating physicians who were trained in quality of life questionnaires and profiles

Exclusion Criteria:

* Secondary breast cancer, patients who refused to participate, patients incapable of filling out questionnaires, male patients, pregnant patients, age below 18 yrs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-11; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
amount of QL-deficits at several intervals and at the end of the study period (1 year postoperatively) | operation till 1 year after operation

CONTACTS AND LOCATIONS:
Overall Officials: Monika KS Klinkhammer-Schalke, MD, Study Chair — Tumor Center Regensburg; Michael MK Koller, Ph.D., Principal Investigator — University of Marburg, Institut of Theoretical Surgery; Brigitte BE Ernst, MD, Principal Investigator — General Practitioner, Bad Abbach; Ferdinand FH Hofstädter, MD, Prof., Principal Investigator — Tumor Center Regensburg; Wilfried WL Lorenz, MD, Prof., Principal Investigator — Tumor Center Regensburg
Locations (1):
- Tumorzentrum Regensburg, Regensburg, Bavaria, Germany

REFERENCES:
- [Background] Koller M, Lorenz W. Quality of life: a deconstruction for clinicians. J R Soc Med. 2002 Oct;95(10):481-8. doi: 10.1177/014107680209501002. No abstract available. PMID 12356967
- See also: Related Info — http://www.tumorzentrum-regensburg.de